CLINICAL TRIAL: NCT00370695
Title: Spinal Cord Stimulation for Chronic and Intractable Back Pain in Patients Who Are Not Surgical Candidates
Brief Title: Spinal Cord Stimulation for Chronic and Intractable Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Data Collected
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCS-03-05
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Back Pain
Keywords: Chronic back pain; Intractable neuropathic back pain; Lumbar radiculopathy; Spinal cord stimulation
MeSH Terms: conditions — Back Pain; Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Precision Spinal Cord Stimulation System (Experimental): Single arm Precision Spinal Cord Stimulation System.
  Interventions: Device: Precision Spinal Cord Stimulation System

INTERVENTIONS:
Device: Precision Spinal Cord Stimulation System — Stimulation turned on from implant throughout the Study

SUMMARY:
The purpose of this study is to evaluate the efficacy of spinal cord stimulation (SCS) using the Precision implantable neurostimulation device for chronic and intractable back pain in subjects who are not candidates for surgery or who have chosen to seek alternative therapy.

DETAILED DESCRIPTION:
Management of symptoms of chronic back pain and/or lumbar radiculopathy is often difficult and inadequate. Current treatment options include pharmacological treatments, physical therapy, nerve blocks, surgical interruption of the pain pathway, or back surgery. Many patients either do not have adequate pain management with conventional treatments or are not able to tolerate the treatments due to significant side effects. Similarly, many patients are either not candidates for surgical interventions, or are unwilling to undergo such procedures. Spinal cord stimulation has proven to be an effective treatment for patients with pain following a failed back surgery, and this study will investigate spinal cord stimulation as a treatment option for the treatment of chronic back pain in patients who have never had back surgery. A successful study outcome will establish spinal cord stimulation as a less-invasive treatment option to be considered prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic and intractable neuropathic back pain and/or lumbar radiculopathy of moderate to severe intensity and have elected Spinal Cord Stimulation (SCS) as next line of treatment.
* Be 18 years of age or older.
* Be an appropriate candidate for the surgical procedures required for SCS implant.
* Be willing and able to comply with all study related procedures and visits.
* Be capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

* Have had any back or spine surgery.
* Have any evidence of neurologic instability or any anatomic problem of the spine that requires surgery.
* Have any other chronic pain conditions likely to confound evaluation of study endpoints.
* Are a current substance abuser (including alcohol and illicit drugs).
* Have a significant psychiatric disorder.
* Have a condition currently requiring or likely to require the use of MRI or diathermy.
* Have an active implantable device.
* Are pregnant or lactating or planning to become pregnant in the next year.
* Have participated in any drug or device trial in the last 4 weeks or plan to participate in any other study during the year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Neuromodulation Corporation
Locations (1):
- Huntley Pain Specialists, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Precision Spinal Cord Stimulation System
Started | 15
12 Weeks Post-activation | 2
Completed | 0
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Precision Spinal Cord Stimulation System
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Study is to Evaluate Back Pain Severity at 12 Weeks Post-activation as Compared to Baseline.
Time Frame: 12 weeks
Population: The study was terminated and efforts were made to locate data. No study data are available.
Arm/Group | Precision Spinal Cord Stimulation System
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through 52 weeks post-activation or withdrawal.
Arm/Group | Precision Spinal Cord Stimulation System
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precision Spinal Cord Stimulation System (N=15)
Popliteal Aneurysm and Clot (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precision Spinal Cord Stimulation System (N=15)
Increased falling (Injury, poisoning and procedural complications) | 1 (1)
Orbital Ecchymosis (Eye disorders) | 1 (1)
Skin tear (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Insufficient data collected to report results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes